CLINICAL TRIAL: NCT00247234
Title: Effectiveness of Group Based Schema Therapy in the Treatment of Borderline Personality Disorder and Avoidant Personality Disorder
Brief Title: Effectiveness of Group Based Schema Therapy in the Treatment of Personality Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ursula.falkmer+AEA-stolav.no
Record Dates: First submitted 2005-10-31; First posted 2005-11-01 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Personality Disorder, Borderline; Avoidant Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder; Personality Disorders | interventions — Schema Therapy; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- schema therapy (Experimental)
  Interventions: Behavioral: Schema Therapy
- standard care (Active Comparator): standard psychiatric out-patient care
  Interventions: Behavioral: standard care

INTERVENTIONS:
Behavioral: Schema Therapy — group based schema therapy
  Arms: schema therapy
Behavioral: standard care — standard psychiatric out-patient care
  Arms: standard care

SUMMARY:
This study intends to compare the effectiveness of schema therapy with standard psychiatric outpatient care for patients with borderline or avoidant personality disorder.

ELIGIBILITY:
Inclusion Criteria:

* Avoidant or Borderline personality disorders

Exclusion Criteria:

* Do not speak Scandinavian languages
* Antisocial personality disorder
* Narcissistic personality disorder
* Affective bipolar disorder I
* Schizophrenia
* Mental impairment/organic brain disorder
* Substance dependence
* Planned pregnancy
* Serious somatic illness
* Anorexia Nervosa

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2004-09 (Actual); Primary Completion 2011-06 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
quality of life | 5 years
  Self-report measures
depression | 5 years
  Self-report measures
anxiety | 5 years
  Self-report measures
suicidal ideation | 5 years
  Self-report measures

SECONDARY OUTCOMES:
Use of psychotropic medication | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Are Holen, M.D., Ph.D., Study Chair — Department of Neuroscience, NTNU - Faculty of Medicine, MTFS, NO-7489 Trondheim, Norway
Locations (1):
- St. Olavs Hospital, Trondheim, Norway